CLINICAL TRIAL: NCT03877471
Title: Safety Study of Human Embryonic Stem Cell Derived Mesenchymal Stem Cell (MSC)-Like Cells Transplantation in Women With Primary Ovarian Insufficiency (POI)
Brief Title: Mesenchymal Stem Cells (MSCs) - Like Cell Transplantation in Women With Primary Ovarian Insufficiency
Acronym: MSCLCTWPOI
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Hongmei Wang, Professor, Chinese Academy of Sciences
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IOZ ChineseAS POI-2
Record Dates: First submitted 2019-03-11; First posted 2019-03-15 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Primary Ovarian Insufficiency
Keywords: Mesenchymal stem cell; Transplantation; Human embryonic stem cell; Premature ovarian failure
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Intervention Model Description: Patients will be subjected into 3 groups, with a low (0.2×107), medium (0.5×107) and high dosage (1.0×107) of cells transplantation for each ovary. The investigator will first carry out the low dosage group, and then the medium dosage group, based on the safety evaluation of the previous group, the high dosage group will be executed in the same way.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dosage (Experimental): The low dosage will inject 2 million MSC-like cells (in 100ul suspension) for each ovary.
  Interventions: Genetic: Cell therapy
- Medium dosage (Experimental): The medium dosage will inject 5 million MSC-like cells (in 100ul suspension) for each ovary.
  Interventions: Genetic: Cell therapy
- High dosage (Experimental): The high dosage will inject 10 million MSC-like cells (in 100ul suspension) for each ovary.
  Interventions: Genetic: Cell therapy

INTERVENTIONS:
Genetic: Cell therapy — Ovary injection with MSC-like cells through transvaginal ultrasound,3 injection points for each ovary.

SUMMARY:
There is a high incidence of women suffering from Primary Ovarian Insufficiency (POI). So far, there was no treatment sufficient enough to cure POI. Cell therapy is a rapidly developing field and have shown immense promise in the treatment of ovarian dysfunction. In this study, the investigator will evaluate the safety of MSC-like cell therapy in women suffering from POI.

DETAILED DESCRIPTION:
The purpose of this work is to explore the safety and preliminary efficacy of human embryonic stem cell derived MSC-like cell transplantation in women with POI. MSC-like cells were injected directly into bilateral ovaries under transvaginal ultrasound. Patients are subjected into 3 groups, with low (0.2×107), medium (0.5×107) and high dosage (1.0×107) of cells injection for each ovary. The outcomes of patients were followed after the injection every 2 weeks. The investigator mainly follow the safety indexes, and the level of sex hormone and signs of follicle growth will also be monitored. The growing follicles will be stimulated by exogenous hormone, followed by oocyte retrieval and in vitro fertilization (IVF).

ELIGIBILITY:
Inclusion Criteria:

1. Under 40 years of age;
2. Have established regular menstrual cycle, oligomenorrhea / amenorrhea ≥ 4 months;
3. FSH (Follicle-Stimulating Hormone) > 25 IU/mL;
4. Bilateral ovaries are visible by ultrasound;
5. Have fertility requirement, husband has sperms;
6. Willing to sign the Informed Consent Form.

Exclusion Criteria:

1. Primary amenorrhea;
2. History of serious drug allergy or allergic constitution;
3. Thrombophlebitis and thromboembolia, past and present;
4. Acute or chronic infection, hematologic disease, angiocardiopathy, pulmonary disease, liver disease, nephropathy, pancreas disease
5. Autoimmune disease, history of severe familial genetic disease, etc.
6. Anatomical abnormality of reproductive system;
7. Contraindications for pregnancy;
8. Spouse azoospermia;
9. HIV+, hepatitis B, C;
10. Thyroid dysfunction;
11. History of previous malignant or ovarian tumors, history of ovarian therapy;
12. Abnormal karyotyping (e.g. turner syndrome, fragile X syndrome);
13. During pregnancy or lactation;
14. Alcohol or other substance abuse;
15. Mental disease, communicate obstruction;
16. Unwilling to comply with follow-up schedule or want to take other treatment during the follow-up period;
17. Attending doctor consider inappropriate to take part in.

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Only female will be enrolled.
Enrollment: 28 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Temperature | 0-24 weeks
  Body temperature of the participants will be measured fortnightly after injection.
Pulse | 0-24 weeks
  Pulse of the participants will be measured fortnightly after injection.
Breaths per minute | 0-24 weeks
  Breathing rate of the participants will be measured fortnightly after injection.
Blood pressure | 0-24 weeks
  Both systolic pressure and diastolic pressure of the participants will be assessed fortnightly after injection.

SECONDARY OUTCOMES:
Number of antral follicle | 0-24 weeks
  The number of antral follicles developing will be recorded by transvaginal ultrasound fortnightly after injection.
Follicle-stimulating hormone (FSH) serum level | 0-24 weeks
  Serum FSH level will be tested fortnightly after injection.
Estradiol (E2) serum level | 0-24 weeks
  Serum E2 level will be tested fortnightly after injection.
Anti-Mullerian hormone (AMH) serum level | 0-24 weeks
  Serum AMH level will be tested fortnightly after injection.
Ovarian volume | 0-24 weeks
  The ovarian volume will be recorded fortnightly by transvaginal ultrasound after injection.

CONTACTS AND LOCATIONS:
Overall Officials: Hongmei Wang, Doctor, Principal Investigator — Institute of Zoology, Chinese Academy of Sciences
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No
The investigator have not recruited enough participant yet, till now, most of them would like to keep the individual participant data classified.